CLINICAL TRIAL: NCT01658618
Title: A Non-Interventional Safety Study Providing 12 Months Follow-up From First Exposure to HP802-247 in Subjects With Venous Leg Ulcer
Brief Title: Safety Study Providing 12 Months Follow-up From First Exposure to HP802-247 in Subjects With Venous Leg Ulcer
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Healthpoint (Industry)
Responsible Party: Sponsor
Other Study IDs: 802-247-09-030
Record Dates: First submitted 2012-08-01; First posted 2012-08-07 (Estimated); Last update posted 2014-02-03 (Estimated); Status verified 2014-01

CONDITIONS: Venous Leg Ulcer
Keywords: Venous leg ulcer; ulcer; venous stasis; compression; venous; venous stasis ulcer; vlu; hp802-247-09-029
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: HP802-247

SUMMARY:
This observations safety study is intended for subject who participated in the 802-247-09-029 study with the investigational product HP802-247 for venous leg ulcers and received at least one application of HP802-247 or Vehicle (an inactive substance). This study is being done for the following purposes:

1. to identify new adverse events,
2. to examine ongoing adverse events not resolved in subjects who participated in the 802-247-09-029 trial,
3. to record wound status, and
4. to determine if there are differences in Health Related Quality of Life (HRQoL) associated with the treatment assignment from the 802-247-09-029 Trial.

Investigational means that HP802-247 has not been approved by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
Inclusion Criteria:

* Provide informed consent document
* Subject was randomized in 802-247-09-029 and received at least one application of a test article.
* Subject has ended their participation in 802-247-09-029 by virtue of completing the study, or by dropping out prior to completion.

Exclusion Criteria:

* Subjects who refuse to provide written informed consent will be excluded from this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohorts will be carried over and include all subjects who were randomized in 802-247-09-029 and received at least one application of a test article. Subjects will be enrolled based on participation in the 802-247-09-029 trial, evidenced by randomization and completion (or discontinuation) in that trial and having received at least one application of test article.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-03 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | 12 months
  The objectives of this study are to identify new adverse events, examine ongoing adverse events not resolved in subjects who participated in the 802-247-09-029 trial, and record wound status.

SECONDARY OUTCOMES:
Exploratory Objectives | 12 Months
  The Health Economic objective for this study is to determine if there are differences in Health related Quality of Life (HRQoL) associated with the treatment assignment from the 802-247-09-029 Trial.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Chair — Chief Medical Officer; Tommy Lee, MSHS, Study Director — Associate Director Clinical Operations; Robert Kirsner, MD, Principal Investigator — Investigator; William Marston, MD, Principal Investigator — Investigator
Locations (44):
- United States (39):
  - Glendale, Arizona
  - Phoenix, Arizona
  - Tucson, Arizona
  - Carlsbad, California
  - Castro Valley, California
  - Laguna Hills, California
  - Long Beach, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Stockton, California
  - Sylmar, California
  - Washington D.C., District of Columbia
  - Gainesville, Florida
  - Hialeah, Florida
  - Miami, Florida
  - South Miami, Florida
  - Tamarac, Florida
  - Chicago, Illinois
  - Jacksonville, Illinois
  - North Chicago, Illinois
  - Springfield, Illinois
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Cambridge, Massachusetts
  - Las Vegas, Nevada
  - Emerson, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Akron, Ohio
  - Tulsa, Oklahoma
  - Dunmore, Pennsylvania
  - Wyomissing, Pennsylvania
  - Dallas, Texas
  - Fort Worth, Texas
  - San Antonio, Texas
  - St. George, Utah
  - Roanoke, Virginia
  - Tacoma, Washington
- Canada (5):
  - Vancouver, British Columbia
  - Greater Sudbury, Ontario
  - Hamilton, Ontario
  - London, Ontario
  - Sherbrooke, Quebec